CLINICAL TRIAL: NCT07154940
Title: Diagnostic Yeild of Esophagogastrodudenoscopy in Pediatric Chronic Abdominal Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amal Ayoub Ibrahim Hinnawi, Resident doctor, Assiut University
Other Study IDs: AUCH AssiutU
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-04

CONDITIONS: Endoscopy in Chronic Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the diagnostic yeild of esophagogastrodudenoscopy in children with chronic abdominal pain

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 18 years presenting with chronic abdominal pain which defined according to the Rome IV criteria as persistent or recurring abdominal pain that has been present for at least 3 months, with symptom onset at least 6 months prior to diagnosis. This pain must be continuous or nearly continuous, and only occasionally related to physiological events like eating or defecation. Furthermore, the pain must limit some aspect of daily functioning, and it is not feigned or explained by another medical condition and referred to GIT unit for Esophagogastroduodenoscopy and not undertreatment based on clinical judgment due to the presence of one or more of the following:

  * Alarm symptoms (e.g., weight loss, anemia, Hematemesis, Dysphagia, persistent vomiting, nocturnal pain)
  * Failure of empiric therapy (e.g., proton pump inhibitors or dietary modifications)
  * Suspicion of an underlying organic disease (e.g., celiac disease or Helicobacter pylori infection)

Exclusion criteria:

1. Acute abdominal pain
2. Children aged less than 6 years and more than 18 years
3. Recent use of proton pump inhibitors (within 2 weeks) or antibiotics (within 4 weeks) before endoscopy.
4. Children meeting the criteria of functional abdominal pain according to Rome IV criteria in which was defined as as recurrent or chronic abdominal pain that is not explained by another medical condition and is not solely associated with physiological events like eating or menstruation. It must occur at least 4 times per month for at least 2 months, and diagnostic evaluation should rule out other conditions .
5. Children with contraindications to undergoing EGD (e.g., severe respiratory or cardiac conditions).
6. Children who refuse to participate or whose parents do not provide consent.
7. Children previously diagnosed with recurrent abdominal pain -

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with chronic abdominal pain
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence of endoscopic and histopathological abnormalities in symptomatic children undergoing esophagogastrodudenoscopy for chronic abdominal pain | Oct 2025 to april 2027

IPD SHARING:
Plan to Share IPD: No